CLINICAL TRIAL: NCT01904942
Title: Study of Hepatocellular Carcinoma in Cirrhotic Patients
Acronym: CIRCE ProSpec
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DUCOROY PHRC K 2010
Record Dates: First submitted 2013-06-26; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The project is based on a case-control study including cirrhotic patients with (200 cases) and without (400 controls) Hepatocellular carcinoma. The determination of sample sizes in proteomic or spectroscopic studies has to be adapted to the high dimensional setting. The proteomic analysis will be conducted by Clinical Innovation Proteomic Platform of Dijon. Two approaches will be used in the proteomic study: A global approach based on the comparison of proteomic spectra profiles obtained after mass spectrometry analysis (MALDI-TOF). The particularity of this study with regard to previous studies is : the procedures used to purify the sub proteomes (Five automated methods including depletion fractionation and purification will be applied), the qualification of the generated data with the introduction of quality controls, the high number of samples included in the study. The second approach BIA-MS (Biomolecular interaction analysis mass spectrometry) is targeted approach allows the capture, quantification and characterization of proteins.

The quality controls allow to quantify the various variability sources and to validate that biological variability is higher than technical variability. All the samples will be treated and analyzed with the same protocols, 100 samples will be used to validate the marker and statistical models developed after analysis of the first 500 samples. The infra-red spectroscopy analysis will be conducted by MéDIAN team, CNRS UMR 6237 of Reims university. The first 300 samples after feature selection reference spectra, are classified into different classes by means of mathematical classification methods such as multivariate statistical processes of pattern recognition, neuronal networks, support vector machines and methods of case-based classification or machine learning, genetic algorithms or methods of evolutionary programming. The analysis of a second set of samples (300) will validate the different mathematical classification methods developed.

In the global study the investigators will unravel the relationship between proteomic, spectroscopic and metabolic/nutritional data. The description of these relationships will use canonical analysis and multi-block analysis in a more general extent. The goal of these methods is to explore relationships that may exist between several groups of quantitative variables observed on the same set of individuals.

ELIGIBILITY:
Inclusion Criteria:

* Cases and controls will be males aged 35 or older, and will give an informed consent to participate in the study. All HCC cases evolving in cirrhotic liver, whatever the etiology of cirrhosis, will be included. Criteria for the diagnosis of HCC will be those defined by the European Association for Study of the Liver (EASL) (Bruix J, J Hepatol 2001): All patients with cirrhosis, whatever its etiology, will be included. The diagnosis of cirrhosis will rely on histological confirmation by liver biopsy:
* In patients free of portal thrombosis at Doppler imaging, on the presence of portal hypertension ascertained by biological (tricytopenia), morphologic (abdominal US, CT or MRI), hepatic venous pressure measurement or upper endoscopy (mosaic gastropathy, varices).
* In patients with portal thrombosis, on the presence of portal hypertension associated with:

  * Clinical (hepatomegaly with clinical evidence of hepatocellular failure: spider naevi, palmar erythema, white nails, gynecomastia) or morphological signs of cirrhosis (enlarged liver, nodular surface, sharp lower edge).
  * And/or biological signs of hepatocellular failure (TP<70%, low albuminemia)
  * And/or sinusoidal block assessed by liver venous gradient >18 mm Hg In the present state of knowledge, a fibrotest value at 4 or a fibroscan value > 12,5 kPa Without any other clinical or biological signs will be considered as diagnosis criteria of cirrhosis only for chronic viral C hepatitis. The lack of HCC in cirrhotic patients at inclusion will be assessed through good quality imaging examinations (abdominal US, CT scan or MRI) and AFP below 100 ng/ml.

Exclusion Criteria:

* - patients under 35years old or more than 75 years of age
* other cancer in evolution
* HIV infection
* major somatic or psychiatric illness not compatible with the inclusion in the study
* non HCC primary liver cancer.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Proteomic investigations | at the baseline

SECONDARY OUTCOMES:
Infrared spectroscopic investigations | at the baseline

CONTACTS AND LOCATIONS:
Overall Officials: DUCOROY Patrick, Principal Investigator — Pole de recherche clinique / CLIPP (Clinical Innovation ProteomicPlatform)